CLINICAL TRIAL: NCT00858884
Title: Libman-Sacks Endocarditis as a Cause of Neuropsychiatric Systemic Lupus Erythematosus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HRRC# 06-117
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2013-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Libman-Sacks endocarditis; Stroke; Transient ischemic attack; Neuropsychiatric systemic lupus erythematosus; Transesophageal echocardiography; Magnetic resonance imaging
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Stroke; Ischemic Attack, Transient; Lupus Vasculitis, Central Nervous System | interventions — Laboratories

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- No intevention (No Intervention): No intervention
  Interventions: Other: Clinical and laboratory evaluations, transesophageal echocardiography, carotid duplex, transcranial duplex, and magnetic resonance of the brain

INTERVENTIONS:
Other: Clinical and laboratory evaluations, transesophageal echocardiography, carotid duplex, transcranial duplex, and magnetic resonance of the brain — All participating subjects (patients with and without neuropsychiatric SLE and healthy controls) will undergo clinical and laboratory evaluations, transesophageal echocardiography, carotid duplex, transcranial duplex, and magnetic resonance of the brain
  Other Names: Clinical and laboratory and imaging tests

SUMMARY:
The purpose of this study is to determine whether Libman-Sacks endocarditis (inflammation of the heart valves) is the cause of neuropsychiatric manifestations (stroke, transient ischemic attacks, cognitive dysfunction, seizures, acute confusional state, or psychosis) in patients with systemic lupus erythematosus.

Hypothesis of the study: Libman-Sacks endocarditis (especially valve vegetations or "small valve growths") generate macro (large) and micro (tiny) emboli that occlude the medium and small cerebral vessels resulting in altered perfusion, ischemic brain injury, and major NPSLE (stroke, TIA, seizures, cognitive dysfunction, acute confusional state, or psychosis).

DETAILED DESCRIPTION:
Specific Aim 1: To determine cross-sectionally in SLE subjects the effects of valve vegetations detected by TEE on the presence of active cerebral microemboli, altered perfusion, ischemic brain lesions, and NPSLE. Findings in SLE patients will be compared to those in controls.

Specific Aim 2: To determine longitudinally in patients with new or recurrent NPSLE and during remission whether valve vegetations, active cerebral microemboli, and abnormal cerebral perfusion improve, or normalize when compared to baseline data in patients without NPSLE or matched controls.

Specific Aim 3: To determine cross-sectionally in SLE subjects the presence of active cerebral microemboli, altered brain perfusion, brain injury, and NPSLE in relation to other valve abnormalities, such as valve thickening or valve regurgitation, in addition to or independently of valve vegetations; and to determine longitudinally these relationships in patients with NPSLE. Findings in SLE patients will be compared to baseline data in patients without NPSLE or matched controls.

Our SLE/NPSLE cohort of >400 subjects and our extensive cardiac and neuroimaging experience with TEE and MR-based techniques are essential resources for this study. We will integrate inflammatory and hemostatic parameters with multiple imaging modalities to investigate the causal connection between valve vegetations and the generation of microemboli and perfusion abnormalities, which then result in brain injury and NPSLE. A causal connection of valve vegetations to brain injury and NPSLE would result in a fundamental shift in the understanding of the pathogenesis, diagnosis, and therapy of Libman-Sacks endocarditis and NPSLE. These findings may extend to other inflammatory diseases associated with valve disease and complicated with central nervous system disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of SLE according to the American Rheumatology Association independent of gender or ethnicity and recruited from the Rheumatology Clinics at the University of New Mexico Health Sciences Center
* Patients (> 18 and < 60 years old) with new or recurrent major NPSLE
* Healthy volunteers based on history and physical examination
* Because of conscious sedation and the MR aspects of the study, women of childbearing potential who agree to participate will require to be on contraception therapy, had undergone an sterilization procedure, or have a negative pregnancy test for their inclusion in the study.

Exclusion Criteria:

* Children (as defined by NIH) will be excluded because the neurocognitive tests are standardized for individuals 18 or older. In New Mexico, adulthood is legally defined as 18 years old. Therefore, inclusion of subjects <18 years old would invalidate the results of neurocognitive testing. Moreover, the number of children below 18 with SLE is so low in our population as to not provide a statistically viable result.
* Subjects older than 60 years will also be excluded because their high prevalence and incidence of aging related valve and brain pathology and neurocognitive dysfunction.
* Pregnant women will not be studied because of the need of conscious sedation during TEE and the MR aspects of the study. Women of childbearing potential who agree to participate and are not on contraception therapy or have not undergone an sterilization procedure will require a negative pregnancy test before their inclusion in the study.
* Patients with known or suspected valve or cardiac disease unrelated to SLE such as rheumatic valve disease, active or healed infective endocarditis, congenital bicuspid aortic valves, myxomatous mitral valves with prolapse, and those with prosthetic valves and/or sustained atrial fibrillation or flutter will be excluded.
* Patients with a known cardiac substrate for embolism (LV or LA thrombi, LV aneurysm, LV ejection fraction <40% will be excluded on enrollment, but the development of these complications during the study will be noted and considered as a separate variable.
* Patients with non-SLE related cardiovascular or CNS disease such as congenital hypercoagulability syndromes, hypertensive encephalopathy, CNS infection, metabolic disturbances, hepatic failure, uncontrolled diabetes, or patients who are medicated with neuroleptic drugs.
* Patients with serious medical illness unsuitable for undergoing TEE and MRI scanning.
* Patients with thrombotic thrombocytopenic purpura (TTP).
* Patients with contraindications to esophageal intubation (i.e. esophageal stricture or esophageal varices).
* Patients at risk for hazard due to magnetic fields will be excluded. In critically ill patients TEE will be postponed until medically stable. Patients with supratherapeutic INR (>3.5) will not undergo TEE until INR <3.5. 11)
* Patients without NPSLE on warfarin at the entry phase of the study.
* History of head trauma in the form of concussion or contusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine cross-sectionally in SLE subjects the effects of valve vegetations on the presence of active cerebral microemboli, altered perfusion, ischemic brain lesions, and NPSLE. Findings in patients will be compared to those in controls. | 4 years

SECONDARY OUTCOMES:
To determine longitudinally in patients with new or recurrent NPSLE if during remission vegetations, cerebral microemboli, and abnormal cerebral perfusion improve, or normalize as compared to baseline data in patients without NPSLE or matched controls. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Roldan, M.D., Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Roldan CA. Valvular and coronary heart disease in systemic inflammatory diseases: Systemic Disorders in heart disease. Heart. 2008 Aug;94(8):1089-101. doi: 10.1136/hrt.2007.132787. No abstract available. PMID 18625800
- [Background] Roldan CA, Qualls CR, Sopko KS, Sibbitt WL Jr. Transthoracic versus transesophageal echocardiography for detection of Libman-Sacks endocarditis: a randomized controlled study. J Rheumatol. 2008 Feb;35(2):224-9. Epub 2007 Dec 15. PMID 18085739
- [Background] Roldan CA, Gelgand EA, Qualls CR, Sibbitt WL Jr. Valvular heart disease by transthoracic echocardiography is associated with focal brain injury and central neuropsychiatric systemic lupus erythematosus. Cardiology. 2007;108(4):331-7. doi: 10.1159/000099104. Epub 2007 Feb 12. PMID 17299260
- [Background] Roldan CA, Gelgand EA, Qualls CR, Sibbitt WL Jr. Valvular heart disease is associated with nonfocal neuropsychiatric systemic lupus erythematosus. J Clin Rheumatol. 2006 Feb;12(1):3-10. doi: 10.1097/01.rhu.0000200378.42836.7f. PMID 16484873
- [Background] Roldan CA, Gelgand EA, Qualls CR, Sibbitt WL Jr. Valvular heart disease as a cause of cerebrovascular disease in patients with systemic lupus erythematosus. Am J Cardiol. 2005 Jun 15;95(12):1441-7. doi: 10.1016/j.amjcard.2005.02.010. PMID 15950567
- [Background] Roldan CA. Valvular disease associated with systemic illness. Cardiol Clin. 1998 Aug;16(3):531-50. doi: 10.1016/s0733-8651(05)70030-8. PMID 9742329
- [Background] Roldan CA, Shively BK, Crawford MH. An echocardiographic study of valvular heart disease associated with systemic lupus erythematosus. N Engl J Med. 1996 Nov 7;335(19):1424-30. doi: 10.1056/NEJM199611073351903. PMID 8875919
- [Background] Roldan CA, Shively BK, Lau CC, Gurule FT, Smith EA, Crawford MH. Systemic lupus erythematosus valve disease by transesophageal echocardiography and the role of antiphospholipid antibodies. J Am Coll Cardiol. 1992 Nov 1;20(5):1127-34. doi: 10.1016/0735-1097(92)90368-w. PMID 1341885
- [Background] Sibbitt WL Jr, Schmidt PJ, Hart BL, Brooks WM. Fluid Attenuated Inversion Recovery (FLAIR) imaging in neuropsychiatric systemic lupus erythematosus. J Rheumatol. 2003 Sep;30(9):1983-9. PMID 12966602
- [Background] Sibbitt WL Jr, Brandt JR, Johnson CR, Maldonado ME, Patel SR, Ford CC, Bankhurst AD, Brooks WM. The incidence and prevalence of neuropsychiatric syndromes in pediatric onset systemic lupus erythematosus. J Rheumatol. 2002 Jul;29(7):1536-42. PMID 12136916
- [Background] Sibbitt WL Jr, Sibbitt RR, Brooks WM. Neuroimaging in neuropsychiatric systemic lupus erythematosus. Arthritis Rheum. 1999 Oct;42(10):2026-38. doi: 10.1002/1529-0131(199910)42:103.0.CO;2-J. No abstract available. PMID 10524673
- [Background] Sibbitt WL Jr, Jung RE, Brooks WM. Neuropsychiatric systemic lupus erythematosus. Compr Ther. 1999 Apr;25(4):198-208. doi: 10.1007/BF02889620. PMID 10349089
- [Background] Sibbitt WL Jr, Haseler LJ, Griffey RR, Friedman SD, Brooks WM. Neurometabolism of active neuropsychiatric lupus determined with proton MR spectroscopy. AJNR Am J Neuroradiol. 1997 Aug;18(7):1271-7. PMID 9282854
- [Derived] Roldan CA, Joson J, Qualls CR, Sharrar J, Sibbitt WL Jr. Premature aortic stiffness in systemic lupus erythematosus by transesophageal echocardiography. Lupus. 2010 Dec;19(14):1599-605. doi: 10.1177/0961203310377088. Epub 2010 Sep 2. PMID 20813797